CLINICAL TRIAL: NCT02963714
Title: Immunogenicity and Persistence of Intramuscular High Dose Recombinant Hepatitis B Vaccine in Hemodialysis Patients in China: a Multicenter Randomized Controlled Trial
Brief Title: Immunogenicity of Hepatitis B Vaccination in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suping Wang (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor-Investigator, Suping Wang, Professor, Shanxi Medical University
Organization: Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012ZX10002001003004001
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B, Vaccine; Randomized Controlled Trial; Hemodialysis; Immunogenicity
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 µg dose hepatitis B vaccine (Experimental): 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 60 µg dose hepatitis B vaccine
- 20 µg dose hepatitis B vaccine (Experimental): 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 20 µg dose hepatitis B vaccine

INTERVENTIONS:
Biological: 60 µg dose hepatitis B vaccine — three-dose, 60 µg per dose
  Arms: 60 µg dose hepatitis B vaccine
Biological: 20 µg dose hepatitis B vaccine — three-dose, 20 µg per dose
  Arms: 20 µg dose hepatitis B vaccine

SUMMARY:
Intramuscular injection of 40 μg hepatitis B vaccine in a standard three-dose schedule or a four-dose schedule is recommended for hemodialysis patients. However, seroconversion rates are inadequate and persistence of immunity remains a challenge.

This is a randomized, controlled trial. The study will evaluate the immunogenicity, immune persistence, and safety of 20 µg and 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6 in hemodialysis patients.

DETAILED DESCRIPTION:
Participants are randomized in a ratio of 1:1 into 20 µg recombinant hepatitis B vaccine group or 60µg recombinant hepatitis B vaccine group.The 20 µg group will receive three intramuscular injections of the 20 µg recombinant hepatitis B vaccine, while the 60 µg group will receive three intramuscular injections of the 60 µg dose at months 0, 1 and 6, respectively. HBsAg and anti-HBs will be tested during the study period. Adverse reactions will be recorded after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Having end-stage renal disease (ESRD) on maintenance hemodialysis
* Aged between 18 and 70 years at enrollment
* Serologically negative for hepatitis B surface antigen (HBsAg) and hepatitis B surface antibody (anti-HBs) at enrollment
* Willing to adhere to the study protocol

Exclusion Criteria:

* Being pregnant
* Acute cytolysis in the last three months before enrollment
* Any vaccination during the month preceding enrollment
* Intolerance or allergy to any component of the vaccine
* Ongoing opportunistic infection
* Hepatitis C virus infection
* Hematological disorder
* Cancer
* Unexplained fever the week before enrollment
* Immunosuppressive or immunomodulating treatment in the last six months
* Renal transplantation or upcoming renal transplantation
* Liver disease
* Other immunocompromised condition not related to ESRD
* An expected survival of < 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, Principal Investigator — Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng Y, Shi X, Shi J, Gao L, Liu G, Cheng Y, Pan M, Li C, Wang J, Guo X, Zhang Y, Liang X, Wang S. Immunogenicity, antibody persistence, and safety of the 60 mug hepatitis B vaccine in hemodialysis patients: a multicenter, randomized, double-blind, parallel-controlled trial. Expert Rev Vaccines. 2017 Oct;16(10):1045-1052. doi: 10.1080/14760584.2017.1367667. Epub 2017 Aug 21. PMID 28803502

RESULTS

PARTICIPANT FLOW:
Groups:
- IM 20μg Group: Participants received 3 intramuscular injections of 20 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
- IM 60μg Group: Participants received 3 intramuscular injections of 60 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
Period: Overall Study
Arm/Group | IM 20μg Group | IM 60μg Group
Started | 176 | 176
Completed | 126 | 126
Not Completed | 50 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM 20μg Group | IM 60μg Group | Total
Number analyzed (Participants) | 176 | 176 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.2) | 45.5 (12.0) | 44.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 88 | 164
  Male | 100 | 88 | 188
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han ethnicity | 176 | 175 | 351
  Hui ethnicity | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  China: Urban | 89 | 101 | 190
  China: Rural | 87 | 75 | 162

OUTCOME MEASURES:

1. Primary Outcome: Anti-HBs Seroconversion Rate at Month 7
Time Frame: Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 141 | 143
Participants | 118 | 132

2. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 42
Time Frame: Month 42
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 109 | 102
Participants | 33 | 40

3. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 36
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 115 | 106
Participants | 41 | 51

4. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 30
Time Frame: Month 30
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 118 | 108
Participants | 48 | 62

5. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 24
Time Frame: Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 120 | 118
Participants | 54 | 78

6. Secondary Outcome: Anti-HBs Concentration at Month 7
Description: Anti-HBs concentration at month 7 as measured by CMIA
Time Frame: Month 7
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 141 | 143
mIU/mL | 1488.5 [1053.7 to 1923.4] | 1916.6 [1413.7 to 2419.4]

7. Secondary Outcome: Anti-HBs Concentration at Month 12
Description: Anti-HBs concentration at month 12 as measured by CMIA
Time Frame: Month 12
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 126 | 126
mIU/mL | 407.8 [227.0 to 588.7] | 476.2 [290.3 to 662.1]

8. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 12
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 126 | 126
Participants | 109 | 114

9. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 7 days after vaccination with the hepatitis B vaccine
Time Frame: Within 7 days after the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 174 | 175
Participants | 14 | 14

10. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 28 days after vaccination with the hepatitis B vaccine
Time Frame: Within 28 days after the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 174 | 175
Participants | 7 | 8

11. Secondary Outcome: Anti-HBs Seroconversion Rate at Month 18
Time Frame: Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 127 | 126
Participants | 77 | 96

12. Other Pre Specified Outcome: High-level Response Rate at Month 7
Time Frame: Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 141 | 143
Participants | 88 | 107

13. Other Pre Specified Outcome: High-level Response Rate at Month 12
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 126 | 126
Participants | 67 | 82

14. Other Pre Specified Outcome: High-level Response Rate at Month 18
Time Frame: Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 127 | 126
Participants | 30 | 38

15. Other Pre Specified Outcome: High-level Response Rate at Month 30
Time Frame: Month 30
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 118 | 108
Participants | 15 | 19

16. Other Pre Specified Outcome: High-level Response Rate at Month 36
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 115 | 106
Participants | 14 | 14

17. Other Pre Specified Outcome: High-level Response Rate at Month 42
Time Frame: Month 42
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 109 | 102
Participants | 8 | 10

18. Other Pre Specified Outcome: High-level Response Rate at Month 24
Time Frame: Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 120 | 118
Participants | 19 | 23

ADVERSE EVENTS:
Arm/Group | IM 20μg Group | IM 60μg Group
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/175
Other Adverse Events (participants affected / at risk) | 8/174 | 8/175
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IM 20μg Group (N=174) | IM 60μg Group (N=175)
pain (Musculoskeletal and connective tissue disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No